CLINICAL TRIAL: NCT05166213
Title: Patients' Attitudes Towards Open-Label Placebo Implementation Into Clinical Practice
Acronym: PATOLP
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02304; ex21Frey
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Open-label Placebos
Keywords: focus group discussions (FGD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Chronic back pain
  Interventions: Other: focus group discussions (FGD)
- Clinically significant menopausal complaints
  Interventions: Other: focus group discussions (FGD)
- Parkinson's disease
  Interventions: Other: focus group discussions (FGD)
- Migraine
  Interventions: Other: focus group discussions (FGD)
- Cancer-related emesis/nausea
  Interventions: Other: focus group discussions (FGD)

INTERVENTIONS:
Other: focus group discussions (FGD) — FGD to explore patients' attitudes/ concerns towards OLP implementation into clinical practice by means of assessment of qualitative information: 1) Patients' attitudes towards clinical usage of OLPs 2) Personal acceptance of OLP intervention 3) Perceived ideas, concerns regarding OLP implementation. Core questions: 1) Attitudes: After all that I told you about placebos, i.e. that there is a concept that patients are openly elucidated that they receive placebos: What does this elicit in you/What is your opinion on this? How do you like the idea? 2) Context of Acceptance: Under which conditions would you personally take placebos knowing that they are placebos? 3) Concerns: Why would you not take openly administered placebos? 4) Ideas for clinical implication: How could an open placebo intervention look like in the hospital? Where could it be possible to receive placebos and how could a placebo intervention in the best manner take place? What would be important from your point of view?

SUMMARY:
The aim of this project is to assess patients' opinions, attitudes, and ideas regarding the administration of OLPs in clinical practice, although they might never have had contact to placebos. A qualitative approach is used and online focus group discussions (FGD) with patients with different clinical conditions, entailing chronic back pain, Parkinson's disease, chronic migraine, chemotherapy induced emesis, and menopausal complaints are conducted.

DETAILED DESCRIPTION:
Substantial placebo effects have been known for several decades for a multitude of physical as well as psychological complaints. It is essential to test the acceptability of Open-label placebos (OLPs) of patients and health professionals. The aim of this project is to assess patients' opinions, attitudes, and ideas regarding the administration of OLPs in clinical practice, although they might never have had contact to placebos. A qualitative approach is used and online focus group discussions (FGD) with patients with different clinical conditions, entailing chronic back pain, Parkinson's disease, chronic migraine, chemotherapy induced emesis, and menopausal complaints are conducted. A semi-structured topic guide with open-ended questions will be used.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed Consent form (see Appendix)
* Capable of consent (language/cognitive)
* At least 18 years of age
* Ability to attend an online conference in regard of physical and psychological condition and technical knowhow and equipment
* In addition, participants have to be affected by one of the following conditions/disorders:

  * Chronic back pain
  * Chemotherapy-induced emesis (last occurrence at least before 14 days and at maximum before one year)
  * Chronic migraine
  * Parkinson's disease
  * Clinically significant menopausal complaints

Exclusion Criteria:

* Severe ailment and medication side-effects which would interfere with study participation (e.g., due to concentration impairment)
* Acute psychological crisis which would affect study participation essentially or suicidality
* Co-morbidity that overlaps in symptoms with the symptoms necessary for inclusion
* Essential psychiatric disorders other than moderate depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited with help of physicians from the following clinics:
  University Hospital Basel Anästhesiologie: Schmerzmedizin Frauenklinik: Gynäkologische Sozialmedizin und Psychosomatik Neurologie: Migräne und Morbus Parkinson Sprechstunden Onkologie und Psychoonkologie Privatklinik Hohenegg AG. Interested patients will receive a flyer of the study and will be asked if they prefer to enter in contact with the study team by themselves or if the study team is allowed to call the patient.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Qualitative data analysis | one time assessment at baseline with a duration from max. 60 minutes.
  Qualitative data analysis using the approach of "Thematic Analysis". This approach helps to identify, analyze, and interpret patterns of meanings in the form of upcoming "themes" in the qualitative data. Important "themes" deriving from the group discussion between the respective patient groups are explored. . In this manner, important subjective factors of OLP acceptance or non-acceptance can be revealed as well as boundaries of differences within opinions.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Frey Nascimento, Dr., Principal Investigator — University of Basel, Faculty of Psychology, Division of Clinical Psychology and Psychotherapy
Locations (1):
- University of Basel, Faculty of Psychology, Division of Clinical Psychology and Psychotherapy, Basel, Switzerland

REFERENCES:
- [Derived] Frey Nascimento A, Bakis B, Gaab J, Schneider T, Papadopoulou A, Ritter M, Bernstein MH, Blease CR, Locher C. Talking placebo: a qualitative study of patients' attitudes toward open-label placebo implementation into clinical practice. Front Psychol. 2025 Jul 31;16:1533663. doi: 10.3389/fpsyg.2025.1533663. eCollection 2025. PMID 40823423